CLINICAL TRIAL: NCT05264610
Title: Retrospective Analysis of the Effects of Perioperative Osteoanabolic Treatment on Patients With Spinal (Fusion) Surgery.
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01201; mu22Rikli2
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Spinal (Fusion) Surgery
Keywords: osteoanabolic treatment; parathyroid hormone (PTH); bone healing disorder
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection (Laboratory tests, Radiologic diagnostics, Patient data taken from existing medical charts) — Data collection: Bone turnover laboratory parameters: alkaline phosphatase (AP), calcium (corrected for albumin), PTH, Calcidiol (25-OH-D3), N-terminales Kollagen Typ 1 -. Propeptid (P1NP), glomerular filtration rate (GFR), calcium/creatinine (in urine); Radiologic diagnostics: Bone densitometry (DEXA), X-rays, computer tomograms, MRI for analysis of time of the bone healing (or a non-union); Patient data taken from existing medical charts: side effects, tolerability of PTH, patient compliance, presence of previous illnesses as risk factors for the formation of pseudoarthrosis, indication for therapy, time at which therapy started and length of therapy with PTH, precise characterization of the operation (type and whether it is a revision or first operation).

SUMMARY:
This study is to review the the effect of PTH on the outcome of spinal fusion surgery by analyzing the procedure with Forsteo (PTH) previously used in the University Hospital Basel and the Endonet Clinic, as part of a retrospective, observational study.

DETAILED DESCRIPTION:
Spinal fusion operations have been performed in patients with risk factors related to healing or bony consolidation. A distinction is made between risk factors that can be influenced, such as nicotine consumption or the intake of glucocorticoids, and non-modifiable risk factors, such as diabetes mellitus or chronic obstructive pulmonary disease (COPD), which impair bone formation. The presence of these risk factors leads to an increased rate of unhealed fusions, which is why ways are being sought to reduce them. One possibility, in addition to correcting the modifiable risk factors, is the use of topical or systemic drugs.

As early as 2009 and 2010, the effect of parathyroid hormone (PTH) on spinal fusions was investigated in animal experiments. In the studies, a significantly better result was found by therapy with PTH.

In 2012, the effect of PTH on the outcome of spinal fusion surgery in post-menopausal women with osteoporosis in his prospective study was investigated, and another study evaluated the optimal duration of PTH therapy. Overall, the studies to date indicate the benefit of pharmaceutical supplemental therapy. For this reason, it was used on a case-by-case basis in patients undergoing spinal surgery at the University Hospital Basel.

This study is to review the results cited above by analyzing the procedure with Forsteo (PTH) previously used in the University Hospital Basel and the Endonet Clinic, as part of a retrospective, observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spinal (fusion) surgery at the Clinic for Spinal Surgery/ University Hospital Basel
* Perioperative osteo-anabolic therapy between January 1st, 2013 and December 31st, 2018.

Exclusion Criteria:

* Contraindications to PTH therapy
* Patients refusing therapy with PTH

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Clinic for Spinal Surgery/ University Hospital Basel who, in cooperation with the Endonet Clinic Basel, underwent perioperative osteo-anabolic therapy between January 1st, 2013 and December 31st, 2018.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Time of bone healing | one time assessment at baseline
  Time of bone healing is analyzed by radiologic diagnostic, evaluation of patient charts and lab parameter analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Suhm, Prof. Dr. med., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland